CLINICAL TRIAL: NCT04009876
Title: Phase II, Multicenter, Open-label, Non-randomized Study of Neoadjuvant Chemotherapy NALIRINOX (5-FU/LV + Oxaliplatin + Nal-IRI) Followed by Chemoradiotherapy in Patients With Rectal Cancer in a Watch-and-wait Program
Brief Title: A Study to Evaluate a Chemotherapy Treatment Followed by Chemo and Radiotherapy in Patients With Rectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundación de investigación HM (Other)
Collaborators: Syntax for Science, S.L (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM-RE-2017-01
Record Dates: First submitted 2019-07-03; First posted 2019-07-05 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Locally Advanced Rectal Cancer (LARC)
MeSH Terms: interventions — irinotecan sucrosofate; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chemotherapy + Surgery (Experimental): Treatment with 5-FU/LV + Oxaliplatin + nal-IRI for 8 cycles followed by standard chemoradiation (5 weeks) and surgical resection
  Interventions: Drug: nal-IRI; Procedure: Surgical resection; Drug: 5-FU/LV; Drug: Oxaliplatin
- Chemotherapy + Watch-and-wait (Experimental): Treatment with 5-FU/LV + Oxaliplatin + nal-IRI for 8 cycles followed by standard chemoradiation (5 weeks) and "watch-and-wait" surveillance protocol.
  Interventions: Drug: nal-IRI; Other: Watch-and-wait; Drug: 5-FU/LV; Drug: Oxaliplatin

INTERVENTIONS:
Drug: nal-IRI — Treatment with 5-FU/LV + Oxaliplatin + nal-IRI for 8 cycles followed by standard chemoradiation (5 weeks)
Procedure: Surgical resection — Surgical resection of the tumour
  Arms: Chemotherapy + Surgery
Other: Watch-and-wait — No surgery approach
  Arms: Chemotherapy + Watch-and-wait
Drug: 5-FU/LV — Treatment with 5-FU/LV + Oxaliplatin + nal-IRI for 8 cycles followed by standard chemoradiation (5 weeks)
Drug: Oxaliplatin — Treatment with 5-FU/LV + Oxaliplatin + nal-IRI for 8 cycles followed by standard chemoradiation (5 weeks)

SUMMARY:
This is an exploratory, open-label, single arm, non-randomized, multicenter, phase II clinical trial to determine the efficacy and clinical complete response rate in patients with rectal cancer and tumor preoperative evaluation after NAC (Neoadjuvant Chemotherapy) with NALIRINOX (5-FU [fluorouracil)/LV [Leucovorin calcium] + oxaliplatin + nal-IRI [Liposomal Irinotecan]) and chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or females, aged ≥ 18 years.
* Agree to participate and sign voluntary written ICF (Informed Consent Form) before any study specific procedure.
* Patients with confirmed histopathological diagnosis of rectal cancer.
* Patients with locally advanced rectal cancer T3-T4N0M0 or TxN+M0 and selected T2N0M0 candidates to watch & wait program.
* Patients considered for neoadjuvant treatment according to usual clinical practice may also be potential candidates.
* ECOG (Eastern Cooperative Oncology Grou)vperformance status 0 or 1.
* Patients who can receive radiotherapy and chemotherapy.
* No prior or concurrent malignant disease unless in complete remission for more than three years, except for adequately treated in situ carcinoma of the cervix, basal or squamous skin cell carcinoma or in situ transitional bladder cell carcinoma.
* Women of childbearing potential (WOCBP) must have a negative serum pregnancy test before study entry. Both women and men must agree to use a highly effective contraceptive measure throughout the treatment period and for six months after discontinuation of treatment.
* Adequate hematologic function: hemoglobin ≥ 9g/dL; WBC (white blood cell count ) ≥ 4000/mm 3 ; neutrophils ≥ 1.5x10 9 /L; platelets ≥ 100x10 9 /L.
* Adequate hepatic function: total bilirubin ≤ 1.5xULN; ALT / AST (Alanine aminotransferase / Aspartate aminotransferase) ≤ 2.5xULN (Upper Limit of Normality) alkaline phosphatase ≤ 3xULN.
* Adequate renal function: creatinine ≤ 1xULN; creatinine clearance ≥ 60ml/min.
* No peripheral neuropathy (< Grade 2)
* No known history of dihydropyrimidine dehydrogenase deficiency (DPD)

Exclusion Criteria:

* Patients with ECOG performance status ≥ 2.
* Stage I (T1N0M0) or stage IV (TxNxM1) AJCC (American Joint Committee on Cancer) rectal cancer.
* Any illness that the investigator considers will substantially increase the risk if the patient participates in the study.
* Pregnant or breast-feeding woman.
* Chronically active hepatitis B or C virus infection.
* Active uncontrolled infection.
* History, within last year, or presence of unstable angina, myocardial infarction, symptomatic congestive heart failure or asymptomatic left ventricular ejection fraction < 50% (assessed by multiple-gated acquisition scan or equivalent by ultrasound) or clinically significant valvular heart disease.
* Peripheral neuropathy (> Grade 1)
* Known history of dihydropyrimidine dehydrogenase deficiency (DPD)
* Known or suspected reactions to any component of the study medication (5-FU, leucovorin, irinotecan or oxaliplatin) or to components of similar chemical or biologic composition.
* Any phycological, familiar, sociological or geographical condition potentially hampering compliance with the study protocol or follow-up schedule.
* Concurrent participation in any other clinical trial likely to interfere with the therapeutic schedule.
* Patients that had received any previous treatment for their rectal cancer (surgery, chemotherapy or radiotherapy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-10-21 (Actual); Study Completion 2022-10-21 (Actual)

PRIMARY OUTCOMES:
cCR (clinical complete response) rate in LARC ( locally advanced rectal cancer ) patients treated with chemo - chemoradiation. | expected 8 months

SECONDARY OUTCOMES:
Overall survival | Through the study completion (estimated to be 15 months)
Relapse-free survival | Through the study completion (estimated to be 15 months)
Disease-free survival | Through the study completion (estimated to be 15 months)
Percentage of patients that follow the "watch-and-wait" surveillance protocol | Through the study completion (estimated to be 15 months)
Overall toxicity | Through the study completion (estimated to be 15 months)
  acute and late toxicity of neoadjuvant treatment (chemo and chemoradiotherapy) according to the Common Toxicity Criteria (CTC) for adverse events (AE)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Cubillo, MD, Study Director — Director
Locations (4):
- Spain (4):
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital Universitario Madrid Sanchinarro, PAU de Sanchinarro, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario 12 de Octubre, Madrid

IPD SHARING:
Plan to Share IPD: Undecided